CLINICAL TRIAL: NCT02270073
Title: Mindfulness Interventions in Outpatient Cognitive Behavior Therapy in Trainee Therapists: The Process Outcome Mindfulness Effects in Trainees (PrOMET)-Study
Brief Title: The Process Outcome Mindfulness Effects in Trainees (PrOMET)-Study
Acronym: PrOMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: University of Trier (Other); University of Zurich (Other); University of Applied Sciences Esslingen (Unknown)
Responsible Party: Principal Investigator, Johannes Mander, Dr, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA6526/2-1(DFG)
Record Dates: First submitted 2014-10-06; First posted 2014-10-21 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Major Depression; Anxiety Disorder
Keywords: Psychotherapy process; Change mechanisms; Mindfulness; Micro-interventions; Mindfulness interventions; Progressive muscle relaxation
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAU + mindfulness intervention (Experimental): In the first five minutes of each of 25 therapy sessions (duration: about 25 weeks), both patient and therapist perform together the brief intervention with mindfulness elements. Participants sit upright in their chairs in a comfortable position at a distance about one meter from the audio recorder. The text is standardized and spoken by Dr. Thomas Heidenreich. During the exercise, participants are instructed to observe their breathing and body sensations. After completion of the mindfulness intervention, the regular therapy session begins.
  Intervention: Cognitive behavior therapy of trainee therapists
  Interventions: Behavioral: Cognitive behavior therapy of trainee therapists
- TAU + progressive muscle relaxation (Active Comparator): In the first five minutes of each of 25 therapy sessions (duration: about 25 weeks), both patient and therapist perform together a short version of progressive muscle relaxation (PMR). Both patient and therapist sit upright in their chairs in a comfortable position at a distance about one meter from the audio recorder. The PMR text is standardized and spoken by Dr. Thomas Heidenreich. Wording is as similar as possible to the mindfulness interventions.During the exercise, participants are instructed to tense and relax arms, face, body and legs. After completion of PMR, the regular therapy session begins.
  Intervention: Cognitive behavior therapy of trainee therapists
  Interventions: Behavioral: Cognitive behavior therapy of trainee therapists
- Treatment as usual (Other): No specific intervention is conducted at the beginning of therapy sessions. Standard cognitive behavior therapy treatment, based on the individualized case conception of the trainee therapist, is conducted during the whole treatment sessions.
  Intervention: Cognitive behavior therapy of trainee therapists
  Interventions: Behavioral: Cognitive behavior therapy of trainee therapists

INTERVENTIONS:
Behavioral: Cognitive behavior therapy of trainee therapists — In all three treatment arms, trainee therapists perform a cognitive behavior therapy (CBT) under conditions of the German health care system. This treatment is not a manualized intervention, but rather based on individualized treatment plans that have been developed together with expert supervisors during a five session diagnostic stage. Treatment duration is 25 sessions, while on average every fourth is supervized by an CBT expert therapist.

SUMMARY:
Background: Mindfulness has its origins in an Eastern Buddhist tradition that is over 2500 years old and can be defined as a specific form of attention that is non-judgemental, purposeful, and focused on the present moment. It has been well established in cognitive behavior therapy in the last decades, while it has been investigated in manualized group settings. Consequently, the demand to investigate mindfulness under effectiveness conditions in trainee therapists has been highlighted.

Methods/Design: To fill in this research gap, the investigators designed the PrOMET-Study. In this study, the investigators will analyze the effects of brief, audio-tape presented, in-session mindfulness interventions conducted by both trainee therapists and their patients at the beginning of individual therapy sessions in a randomized, controlled longitudinal design under effectiveness conditions in a total of 30 trainee therapists and 150 patients in a large outpatient training center. The investigators hypothesize the mindfulness intervention will have positive effects on therapeutic processes and outcome in contrast to a progressive muscle relaxation and a treatment as usual group. The investigators will conduct multilevel modeling to address the nested data structure.

Discussion: The study results could provide important practical implications, as they could inform ideas on how to improve clinical training of psychotherapists that could be implemented very, as there is no need for complex infrastructures or additional time concerning these brief, in-session mindfulness interventions that are directly implemented in treatment sessions.

DETAILED DESCRIPTION:
Objectives.The main purpose of this study is to identify whether mindfulness exercises carried out at the beginning of individual therapy sessions help to improve the therapeutic process. More specifically, the investigators will examine the effects of a five minute in-session mindfulness intervention practiced by both outpatient and CBT trainee therapist at the beginning of 25 therapy sessions (duration: about 25 weeks) on the processes of therapeutic change measured with a session questionnaire completed after each of these 25 sessions (duration: about 25 weeks) and on clinical outcome assessed every 10 weeks starting at baseline under effectiveness conditions. Thus, before the start of therapeutic treatment, patients are randomized either to a treatment as usual + mindfulness intervention group (TAU+M), a control group practicing a short form of PMR (TAU+PMR), or a treatment as usual (TAU) group. Before the start of the intervention study, all therapists will participate in a six-week workshop-based mindfulness program. The investigators will examine the following hypotheses:

1. The investigators hypothesize that both patients and therapists of the TAU+M will experience higher levels of therapeutic alliance, as represented by the Working Alliance Inventory - Short Revised (WAI-SR), compared to the TAU+PMR and TAU.
2. The investigators hypothesize that in the TAU+M, there will be stronger reductions in clinical symptomatology of patients compared to the TAU+PMR and TAU.

   1. There should be a stronger reduction in clinical symptomatology in the TAU+M versus the TAU+PMR and TAU after the first 25 sessions (duration: about 25 weeks), during which the mindfulness exercise is carried out.
   2. This stronger reduction in clinical symptomatology should remain stable until follow-up.

Methods/Design. The study is a randomized controlled trial with three active treatment arms (TAU+M, TAU+PMR and TAU) under effectiveness conditions.It will be performed at the Center for Psychological Psychotherapy (CPP), a large university outpatient-training center for CBT at the University of Heidelberg. Approximately 1000 patients per year with different types of psychiatric disorders (about two-thirds suffering from anxiety and depression) are treated by approximately 100 trainee therapists there. Patients and therapists of the MIG perform together a brief, five-minute mindfulness exercise at the beginning of 25 therapy sessions (sessions performed on a weekly basis). Patients and therapists of the CG perform together a brief, five-minute version of progressive muscle relaxation at the beginning of 25 therapy sessions. In the TAU group, CPP standard psychotherapy procedure without interventions at the beginning of therapy sessions will be performed. Session-quality assessment will be performed after each of 25 therapy sessions from both patient and therapist perspective. Outcome assessment will be performed at baseline, every ten sessions during treatment, at the end of therapy, and at 12-months follow-up. A detailed description of the outcome measures is to be found under the "Primary and Secondary Outcome" sections.

Participants. A total of 30 trainee therapists and 150 patients will be recruited at the CPP. The general inclusion criterion for patients is a primary depressive or anxiety disorder diagnosis in the Structured Clinical Interview for the Diagnostic and Statistical Manual-IV (DSM-IV), German version. The investigators chose these two disorder groups as patients treated at German university therapy-training centers; approximately 40% suffer from a primary major depression as diagnosed, and approximately 30% suffer from a primary anxiety disorder as diagnosed. Hence, the investigators results will be of importance to a majority of outpatient diagnostic groups. General exclusion criteria for patients will be as follows: (1) an age below 18 or above 59 years, (2) insufficient German language skills, (3) suffering from a psychotic disorder. Other comorbidities are not considered as limitations to entering the study. Power analyses with G*Power and clinical considerations resulted in a sample size of 75 patients with depression and 75 patients with anxiety disorders.

Randomization. A total sample of 150 patients will be assigned to one of the three groups by a stratified randomization process. The randomization process will be performed after a five session diagnostic stage. Patients will be stratified into one of two categories: one group with the main diagnosis of major depression and the other group with the main diagnosis of anxiety disorder. Then, an online randomization will be performed by two independent research assistants.

Mindfulness workshop training. In order to prepare the 30 trainee therapists for the in-session mindfulness interventions outlined in the next section, the investigators will first offer two workshops separated by a six-week home-practice interval to all trainee therapists participating in the study. The workshops will be offered once every year when a new group of trainee therapists starts their outpatient therapies. The first workshop will provide a theoretical background in mindfulness. In the six-week interval between workshops one and two, participants will practice formal and informal mindfulness activities at home. In the second workshop, specifically addressing the mindfulness experiences of participants and suggestions for further improvements will be the focus.

Experimental Session.The experiment will be conducted at the university training center CPP. During the five-minute mindfulness experimental task, both patient and therapist of the TAU+M sit at a distance about one meter from the audio recorder. After the initial greeting ritual, both patient and therapist perform together the brief mindfulness intervention for the first five minutes of the therapy session. While performing the exercise, patient and therapist sit upright in their chairs in a comfortable position, with their feet flat on the floor, arms and legs uncrossed, and hands resting in their laps. The mindfulness text is standardized and spoken by Dr. Thomas Heidenreich, an internationally renowned expert on mindfulness research. During the exercise, participants are instructed to observe their body sensations, followed by non-judgemental and purposeful acknowledgements of personal problems and resources of the patient. After completion of the mindfulness intervention, the regular therapy session begins. Following the treatment session, both patient and therapist complete the session questionnaire described under "Primary and Secondary Outcomes", which requires about two minutes. The TAU+PMR also receives a five-minute audiotaped exercise under basically the same conditions; more specifically, they will receive a short version of PMR that is also spoken by Dr. Heidenreich. On the one hand, PMR is a broadly accepted and easy to implement relaxation exercise that is applied most often as a control intervention when investigating mindfulness interventions. On the other hand, it does not include the hypothesized specific effective ingredients of the mindfulness intervention (mindful observation of physiological and psychological conditions). The wording of the control intervention is as similar to the experimental mindfulness intervention as possible. The TAU will conduct standard individual therapy sessions as usual at the CPP.

Recruitment of patients and therapists. Standard procedure at the CPP is that patients are listed on a waiting list after a diagnostic screening phone call. After patients are listed on the waiting list, they will be contacted by the study team and receive verbal and written information on the study. At the beginning of every year, a group of trainee therapists at the CPP starts their outpatient therapies. Consequently, trainees receive at the beginning of every year verbal and written information on the study. Trainees who participate in the study will then participate in the two mindfulness workshops described above that are offered at the beginning of every year. The information given to the participants of the study includes a precise description of inclusion and exclusion criteria, information concerning the interventions and questionnaires as well as the data collection procedure. Further, it will be emphasized that study participation is on a voluntary basis and that there is the option to revoke consent to participate in the study at any time without having to cite reasons or suffering disadvantages. Moreover, participants have the opportunity to instruct the study team to delete their data without providing reasons.

Development and feasibility of the intervention. The mindfulness exercise was developed in an iterative process in multiple steps: First, Dr. Heidenreich and Dr. Mander phrased a preliminary version based on the breathing space exercise by Michalak, Heidenreich and Williams and on the mindfulness centering exercise by Eifert and Forsyth. Further, 10 therapists and 10 patients conducted this preliminary exercise in one therapy session and delivered feedback. After improving the exercise according to these patient and therapist feedbacks, five mindfulness experts and two experts in psychotherapy process research reviewed the exercise and offered feedbacks for improvement. Based on these feedback processes, the final version of the mindfulness intervention was developed.The feasibility of the brief in-session mindfulness intervention and of the PMR intervention was tested in a pre-study with 12 therapists and 12 patients. Both patients and therapists conducted the exercise at the beginning of one therapy session at the CPP and completed the session questionnaire after the therapy session. Additionally, they completed questions on a scale from 0 (does not apply) to 4 (applies fully) concerning the feasibility of the interventions. The results indicated that the interventions could be integrated without problems in the everyday therapeutic process, that the instructions were understandable and that the exercises generally had a positive impact on the therapy sessions.

Statistical Analysis. The investigators will apply a multilevel modeling approach to address the nested data structure (sessions at level 1 nested within patients at level 2 nested within therapists at level 3): Thereby, the investigators will treat time as a within-subject factor and treatment condition as a between-subject factor. The investigators will analyze main effects, that is, differences in intercepts of TAU+M versus TAU+PMR versus TAU concerning process and outcome variables, and interactive effects, that is, differences in slopes of TAU+M versus TAU+PMR versus TAU concerning process and outcome variables. The investigators statistical hypothesis implies that the intercept is significantly higher in the TAU+M than in the TAU+PMR and the TAU concerning both process and outcome variables. Additionally, it implies that the slope increases significantly stronger in the TAU+M than in the TAU+PMR and the TAU concerning both process and outcome variables. The investigators will conduct analyses on the intention-to-treat sample as well as on the completer sample. Further, patients and therapists pre-treatment characteristics will be investigated as outcome predictors at levels 2 and 3 to control for differential effects on outcome in the three treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* depressive disorder
* anxiety disorder
* treatment at the Center for Psychological Psychotherapy, University of Heidelberg

Exclusion Criteria:

* age below 18 or above 65
* insufficient German language skills
* psychotic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Working Alliance Inventory - Short Revised (WAI-SR) | measured for 25 weeks on weekly basis, starting on first treatment day
  The WAI-SR is a self-report of therapeutic alliance measuring Bond, Goals and Tasks in psychotherapy based on feedback of both patients and therapists concerning the current therapy session
Brief Symptom Inventory (BSI) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Self-report on general symptom severity of patients

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Self-report on depressive symptoms of patients
Inventory of Interpersonal Problems (IIP) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Self-report on interpersonal problems of patients
Kentucky Inventory of Mindfulness Skills (KIMS) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Self-report on patients and therapists mindfulness abilities
Global Assessment of Functioning (GAF) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Therapist perspective on patient´s general symptomatology
Development of Psychotherapists Common Core Questionnaire (DPCCQ) short version | on first treatment day, then on average: 15 weeks, and 12-months follow-up
  Self-report on therapists-variables from therapist perspective
Scale for the Multiperspective Assessment of General Change Mechanisms in Psychotherapy (SACiP) | on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Instrument to assess general therapeutic change mechanisms
Beck Anxiety Inventory (BAI) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Self-report on anxiety symptoms of patients

OTHER OUTCOMES:
Practice Quality-Mindfulness (PQ-M) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks and 12-months follow-up
  Measures presence of therapists and patients during the interventions at beginning of therapy sessions
General Mindfulness Practice (GMP) | on first treatment day, then on average: after 5 weeks, 15 weeks, 25 weeks, and 12-months follow-up
  Instrument to assess therapists personal mindfulness practice, experience before entering study and intensity of mindfulness application in therapy sessions
Therapist Presence Inventory (TPI) | on average: after 5 weeks, 15 weeks, 25 weeks
  Instrument to assess general session presence

CONTACTS AND LOCATIONS:
Overall Officials: Johannes V Mander, PhD, Principal Investigator — Center for Psychological Psychotherapy - University of Heidelberg; Hinrich Bents, PhD, Study Director — Center for Psychological Psychotherapy - University of Heidelberg; Sven Barnow, PhD, Study Chair — Department of Clinical Psychology and Psychotherapy - University of Heidelberg; Christoph Flueckiger, PhD, Study Chair — Department of Clinical Psychology and Psychotherapy - University of Zuerich; Thomas Heidenreich, PhD, Study Chair — Faculty of Social Work, Health and Nursing - University of Applied Sciences Esslingen; Wolfgang Lutz, PhD, Study Chair — Department of Clinical Psychology and Psychotherapy - University of Trier
Locations (1):
- Center for Psychological Psychotherapy - University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Mander J, Kroger P, Heidenreich T, Fluckiger C, Lutz W, Bents H, Barnow S. The Process-Outcome Mindfulness Effects in Trainees (PrOMET) study: protocol of a pragmatic randomized controlled trial. BMC Psychol. 2015 Jul 17;3(1):25. doi: 10.1186/s40359-015-0082-3. eCollection 2015. PMID 26185680
- [Background] Blanck P, Perleth S, Heidenreich T, Kroger P, Ditzen B, Bents H, Mander J. Effects of mindfulness exercises as stand-alone intervention on symptoms of anxiety and depression: Systematic review and meta-analysis. Behav Res Ther. 2018 Mar;102:25-35. doi: 10.1016/j.brat.2017.12.002. Epub 2017 Dec 20. PMID 29291584
- [Background] Mander, J., Kröger, P., Blanck, P., Call, M., Bents, H., & Heidenreich, T. (2017). Theorie- Praxis-Netzwerke in verhaltenstherapeutischer Ausbildung: Schulung, Selbsterfahrung und Einsatz in der Therapie am Beispiel von Achtsamkeit [Theory- Practice Networks for Training in Behavioral Therapy: Training, Self-Discovery and Integration into Treatment Using Mindfulness as an Example]. Verhaltenstherapie, 27(2), 97-106.
- [Result] Mander J, Blanck P, Neubauer AB, Kroger P, Fluckiger C, Lutz W, Barnow S, Bents H, Heidenreich T. Mindfulness and progressive muscle relaxation as standardized session-introduction in individual therapy: A randomized controlled trial. J Clin Psychol. 2019 Jan;75(1):21-45. doi: 10.1002/jclp.22695. Epub 2018 Oct 8. PMID 30295914